CLINICAL TRIAL: NCT04012476
Title: Determination of Parathyroid Function by Fluorescence With Indocyanine Green (ICG) After Total Thyroidectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Son Espases (Other)
Collaborators: Universitat de les Illes Balears (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ICG-Parathyroid
Record Dates: First submitted 2019-06-28; First posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Hypocalcemia; Total Thyroidectomy; Hypoparathyroidism Postprocedural
Keywords: Hypocalcemia post-thyroidectomy; Indocyanine green; Fluorescence guided surgery; Parathyroid fluorescence
MeSH Terms: conditions — Hypocalcemia | interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: Single group: patients undergoing total thyroidectomy with intraoperative infusion of intravenous indocyanine green A prospective unicentric and open clinical trial in which the fluorescence intensity of the parathyroid glands after indocyanine administration will be compared between two groups of patients: those with post-thyroidectomy hypocalcemia and patients who do not present it.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ICG (Experimental): Patients undergoing total thyroidectomy with visualization of the parathyroid glands under infrared light after intraoperative intravenous injection of 5 mg of indocyanine green
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — Administration of 5 mg of intravenous indocyanine green after total thyroidectomy for measurement of parathyroid fluorescence under infrared light
  Other Names: ICG

SUMMARY:
The intensity of parathyroid fluorescence that occurs after intravenous injection of indocyanine green during the performance of a total thyroidectomy correlates with postoperative parathyroid function and could be used as a diagnostic marker of postoperative hypoparathyroidism and hypocalcemia.

DETAILED DESCRIPTION:
The main objective of the study is to compare the intensity of parathyroid fluorescence among patients who present post-thyroidectomy hypocalcemia with that of patients who do not have it. Therefore, the following points will be studied:

* To study the correlation between parathyroid vascularization (intraoperative fluorescence intensity) and postoperative glandular function (serum calcium and parathormone levels).
* To compare the surgeon's subjective assessment of parathyroid fluorescence in the groups of patients with and without postoperative hypocalcemia.
* To compare the objective assessment of parathyroid fluorescence, by using specific computer software developed ad hoc, in the groups of patients with and without postoperative hypocalcemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are going to undergo total thyroidectomy, with or without cervical lymph node dissection.
* Visualization of 2 or more parathyroid glands during the surgical act.
* Normal renal and hepatic functions.
* Absence of a history of hypersensitivity reactions to iodine or indocyanine green.
* Able to understand the nature and protocol of the study and its procedures
* Willingness to participate with the subsequent signing of informed consent.

Exclusion Criteria:

* Age <18 years
* Hepatic or renal insufficiency
* Hypersensitivity to iodine or to indocyanine green.
* Pregnancy or lactation
* Inability to understand the nature and procedures of the study.
* Patients with known preoperative hyperparathyroidism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Calcemia | Day 1 after surgery
  Serum calcium level at 24 hours postoperatively
Subjective parathyroid fluorescence | Intraoperatively
  Fluorescence intensity of the parathyroid glands after administration of indocyanine green (ICG), measured on a subjective analogue scale (0: no fluorescence, 1: hypofluorescence or heterogeneous fluorescence, 2: homogeneous hyperfluorescence).
Objective parathyroid fluorescence | Intraoperatively
  Fluorescence intensity of the parathyroid glands after administration of indocyanine green (ICG), measured by specific computer software developed ad hoc.

SECONDARY OUTCOMES:
Age | Baseline
  Patient's age
Sex | Baseline
  Patient's gender
Body mass index | Baseline
  Patient's BMI
Surgery date | Baseline
  Day when surgery takes place
Preoperative diagnosis | Baseline
  Thyroid pathology indicating total thyroidectomy (thyroid carcinoma, atypical of uncertain significance, goiter or lymphocytic thyroiditis)
Vitamin D | Preoperative blood test
  Preoperative vitamin D level
PTH preop | Immediately before surgery
  Preoperative PTH level
PTH 10 min | 10 minutes post-thyroidectomy
  PTH levels 10 minutes post-thyroidectomy
Surgery | Inmediately after surgery
  Scope of surgery: total thyroidectomy (TT), TT with central neck dissection, or TT with functional lateral neck dissection
Time | Inmediately after surgery
  Duration of surgery
Parathyroid glands | During surgery
  Number of parathyroid glands located during surgery,
Parathyroid gland location | During surgery
  Location of the parathyroid glands (superior right, inf-right, sup-left, inf-left).
Pathologic result | during the first month after surgery
  Outcome of thyroid pathology (papillary carcinoma, nodular hyperplasia or lymphocytic thyroiditis)
Thyroid weight | during the first month after surgery
  Thyroid weight
PG in piece | during the first month after surgery
  Presence of parathyroid glands in the surgical piece and number
Stay | During the first month after surgery
  Number of days of postoperative hospital stay until the day of hospital discharge, measured as full days of 24 hours
Drain | Inmediately after surgery
  Presence and number of surgical drainages
PTH day 1 | Day 1 after surgery
  PTH levels in the postoperative follow-up,
Complications | During the first month after surgery
  Emergence of postoperative complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Son Espases, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vidal Fortuny J, Belfontali V, Sadowski SM, Karenovics W, Guigard S, Triponez F. Parathyroid gland angiography with indocyanine green fluorescence to predict parathyroid function after thyroid surgery. Br J Surg. 2016 Apr;103(5):537-43. doi: 10.1002/bjs.10101. Epub 2016 Feb 11. PMID 26864909
- [Background] Vidal Fortuny J, Sadowski SM, Belfontali V, Guigard S, Poncet A, Ris F, Karenovics W, Triponez F. Randomized clinical trial of intraoperative parathyroid gland angiography with indocyanine green fluorescence predicting parathyroid function after thyroid surgery. Br J Surg. 2018 Mar;105(4):350-357. doi: 10.1002/bjs.10783. Epub 2018 Feb 6. PMID 29405252
- [Background] Lang BH, Wong CK, Hung HT, Wong KP, Mak KL, Au KB. Indocyanine green fluorescence angiography for quantitative evaluation of in situ parathyroid gland perfusion and function after total thyroidectomy. Surgery. 2017 Jan;161(1):87-95. doi: 10.1016/j.surg.2016.03.037. Epub 2016 Nov 10. PMID 27839936
- [Background] Zaidi N, Bucak E, Yazici P, Soundararajan S, Okoh A, Yigitbas H, Dural C, Berber E. The feasibility of indocyanine green fluorescence imaging for identifying and assessing the perfusion of parathyroid glands during total thyroidectomy. J Surg Oncol. 2016 Jun;113(7):775-8. doi: 10.1002/jso.24237. Epub 2016 Apr 4. PMID 27041628
- [Background] Galvez-Pastor S, Torregrosa NM, Rios A, Febrero B, Gonzalez-Costea R, Garcia-Lopez MA, Balsalobre MD, Pastor-Perez P, Moreno P, Vazquez-Rojas JL, Rodriguez JM. Prediction of hypocalcemia after total thyroidectomy using indocyanine green angiography of parathyroid glands: A simple quantitative scoring system. Am J Surg. 2019 Nov;218(5):993-999. doi: 10.1016/j.amjsurg.2018.12.074. Epub 2019 Jan 4. PMID 30665612
- [Background] Rudin AV, McKenzie TJ, Thompson GB, Farley DR, Lyden ML. Evaluation of Parathyroid Glands with Indocyanine Green Fluorescence Angiography After Thyroidectomy. World J Surg. 2019 Jun;43(6):1538-1543. doi: 10.1007/s00268-019-04909-z. PMID 30659346
- [Result] Bonnin-Pascual J, Alvarez-Segurado C, Jimenez-Segovia M, Bianchi A, Bonnin-Pascual F, Molina-Romero FX, Gonzalez-Argente FX. Contributions of fluorescence to endocrine surgery. Cir Esp (Engl Ed). 2018 Nov;96(9):529-536. doi: 10.1016/j.ciresp.2018.09.005. Epub 2018 Oct 14. English, Spanish. PMID 30327136